CLINICAL TRIAL: NCT03726151
Title: Comparative Effectiveness of System Interventions to Increase HPV Vaccine Receipt in FQHCs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of California, Los Angeles (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Roshan Bastani, Professor, Health Policy and Management, UCLA Fielding School of Public Health, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PCS-2017C1-6482
Record Dates: First submitted 2018-10-26; First posted 2018-10-31 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Human Papillomavirus Infection
Keywords: Human Papillomavirus; Immunization; Oncogenic viruses; Cervical Cancer; Health Disparities; Comparative effectiveness; System-level Intervention; Federally Qualified Health Centers
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (No Intervention)
- Parent Reminders (Experimental)
  Interventions: Behavioral: Parent Reminders
- Multicomponent clinic-system strategies (Experimental)
  Interventions: Behavioral: Multicomponent clinic-system strategies
- Combined Condition (Experimental)
  Interventions: Behavioral: Combined Condition

INTERVENTIONS:
Behavioral: Parent Reminders — Automated, system-generated mailed or text message reminders
  Arms: Parent Reminders
Behavioral: Multicomponent clinic-system strategies — 1. Workflow modifications to reduce missed opportunities for vaccination
  2. Provider- and clinic-level audit and feedback
  3. Provider & staff training on workflow modifications and communication strategies
  Arms: Multicomponent clinic-system strategies
Behavioral: Combined Condition — Parent reminders and multicomponent clinic-system strategies
  Arms: Combined Condition

SUMMARY:
UCLA and Northeast Valley Health Center (NEVHC), a large, multi-site Federally Qualified Health Center (FQHC), are partnering to address underutilization of the prophylactic HPV vaccine among underserved, ethnic minority adolescents receiving care through FQHCs. We will use a cluster randomized 2x2 stepped-wedge factorial study design, implemented in seven NEVHC clinics, to compare the effectiveness of parent reminders (mailed and text), multi-component clinic system strategies, a combined intervention (parent reminders + clinic system strategies) and usual care on HPV vaccine series completion among NEVHC adolescent patients. FQHCs provide essential health care to underserved groups and have the infrastructure to sustain effective strategies to improve preventive care delivery. Therefore, study findings will be invaluable for informing future efforts to improve HPV vaccination at the population-level.

DETAILED DESCRIPTION:
The primary aims of this study are to: 1) Examine the effects of two types of parent reminders (mailed, text) and multicomponent clinic system strategies on HPV vaccine completion compared to usual care, 2) Examine the comparative effectiveness of the reminders versus the clinic system strategies and 3) Examine whether combining parent reminders with the clinic system strategies produces larger effects compared to either type of intervention implemented alone.

Additional aims include:

* Explore the relationship between child age (12-14 years versus 15-17 years) and intervention effectiveness, due to the difference in dosing schedules for the two age groups.
* Examine parent (e.g., language preference) and provider (e.g., specialty) characteristics that may act as moderators of intervention effectiveness.
* Assess parent perspectives and experiences related to the different interventions.
* Examine the implementation process (including adaptations) for each of the interventions.
* Disseminate study findings widely to a local and national audience of relevant stakeholders.

The multicomponent clinic system strategies include workflow modifications to minimize missed opportunities for vaccination, provider- and clinic-level audit and feedback, establishment of clinic-level policies and protocols, and will also include provider and staff training regarding workflow modifications and patient communication strategies.

The study will be implemented across six study periods of 12 months each. The seven NEVHC clinics will be randomized into three groups (A, B, C). Following a 12-month start-up and observation period (Period 1), as part of a stepped wedge design, Group A will implement the parent reminders beginning in Period 2, Group B will implement the clinic-based intervention beginning in Period 3, and Group C will implement the combined condition beginning in period 4. In Period 5, Group A will crossover to the combined condition. This change from the original protocol was approved by the study funder as of Fall 2021.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient at one of the seven Northeast Valley Health Corporation (NEVHC) clinics participating in this study
* Has had at least one appointment at NEVHC in the last 2 years
* Must be aged 11-17

Exclusion Criteria:

* Is not a patient at one of the seven Northeast Valley Health Corporation (NEVHC) clinics participating in this study
* Has not had an appointment at NEVHC in the last 2 years
* Is not aged 11-17

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccine series completion based on electronic health record data | 1 year
  We will assess completion of the HPV vaccine series based on the number and the timing of the HPV vaccine doses received according to data in NEVHC's electronic health record system. We will determine completion status based on guidelines from the CDC Advisory Committee on Immunization Practices. For adolescents who initiated the HPV vaccine series before the age of 15, completion will be defined as receiving 2 doses of the HPV vaccine a minimum of 5 months apart. For adolescents who initiated the HPV vaccine series at age 15 or older, completion will be defined as having received 3 doses with the second dose administered at least one month after the first, the third dose received at least 3 months after the second, and the first and third doses administered at least 5 months apart from each other.

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Bastani, PhD, Principal Investigator — Professor, Health Policy and Management, UCLA Fielding School of Public Health; Beth Glenn, PhD, Principal Investigator — Professor, Health Policy and Management, UCLA Fielding School of Public Health
Locations (7):
- United States (7):
  - Northeast Valley Health Corporation- Canoga Park, Canoga Park, California
  - Northeast Valley Health Corporation- Pacoima, Pacoima, California
  - Northeast Valley Health Corporation- San Fernando, San Fernando, California
  - Northeast Valley Health Corporation- Santa Clarita, Santa Clarita, California
  - Northeast Valley Health Corporation- Sun Valley, Sun Valley, California
  - Northeast Valley Health Corporation- Valencia, Valencia, California
  - Northeast Valley Health Corporation- Van Nuys, Van Nuys, California